CLINICAL TRIAL: NCT01526642
Title: Home Non-invasive Ventilation Versus Long-term Oxygen Therapy in COPD Survivors of Acute Hypercapnic Respiratory Failure. A Multicenter Randomized Controlled Trial
Brief Title: Home Non-invasive Ventilation for Chronic Obstructive Pulmonary Disease Patients
Acronym: NIVOLD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/080/HP
Record Dates: First submitted 2012-01-23; First posted 2012-02-06 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Hypercapnic Respiratory Failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Long Term Oxygen Therapy (No Intervention)
- Non Invasive Ventilation (Active Comparator)
  Interventions: Device: Non Invasive Ventilation

INTERVENTIONS:
Device: Non Invasive Ventilation — NIV during night
  Arms: Non Invasive Ventilation

SUMMARY:
Chronic Obstructive Pulmonary disease (COPD) patients with chronic hypercapnic respiratory failure are more likely to develop exacerbations. Non-invasive ventilation has been proposed to treat acute respiratory failure but little information is available about the benefits of home non-invasive ventilation in COPD patients with chronic hypercapnic respiratory failure surviving an acute hypercapnic respiratory failure. The purpose of this study is to determine whether home non-invasive ventilation can reduce recurrent acute hypercapnic respiratory failure in COPD patients who survived an episode of acute hypoxemic respiratory failure (AHRF) treated by Non-invasive ventilation (NIV).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* COPD patients who survived after an episode of acute hypercapnic respiratory failure
* Patients weaned from ventilation (non invasive ventilation or mechanical ventilation) for acute episode since at least seven days with stable arterial blood gas since at least two days: PaCO2 > 55 mmHg and pH > 7.35

Exclusion Criteria:

* Age > 85 years old
* Non- COPD causes of respiratory failure
* Obstructive sleep apnea excluded by polysomnography
* Adverse psychosocial status
* Serious co-morbidity

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Acute hypercapnic respiratory failure episode | up to 102 weeks

SECONDARY OUTCOMES:
Death | 1 month and every 6 months during 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rouen, Rouen, France

REFERENCES:
- [Derived] Lamia B, Cuvelier A, Benichou J, Muir JF. [A multi-centre randomized controlled trial of domiciliary non-invasive ventilation vs long-term oxygen therapy in survivors of acute hypercapnic respiratory failure due to COPD. Non-invasive ventilation in obstructive lung disease (NIVOLD) study]. Rev Mal Respir. 2012 Nov;29(9):1141-8. doi: 10.1016/j.rmr.2012.09.006. Epub 2012 Oct 16. French. PMID 23200590